CLINICAL TRIAL: NCT02401633
Title: A Randomized Trial Comparing the Effect of a Simplified Form of Cardiopulmonary Resuscitation (CPR) Consisting of Only Chest Compressions Compared to CPR With Compressions and Rescue Breaths - the PILOT
Brief Title: Compression Only-CPR Versus Standard-CPR
Acronym: TANGO2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Swedish Heart Lung Foundation (Other)
Responsible Party: Principal Investigator, Jacob Hollenberg, MD, PhD, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCT
Record Dates: First submitted 2015-03-07; First posted 2015-03-30 (Estimated); Last update posted 2022-09-19 (Actual); Status verified 2022-09

CONDITIONS: Cardiac Arrest; Out of Hospital Cardiac Arrest
Keywords: Cardio-Pulmonary-Resuscitation; Advanced Cardiac Life Support; Compression-Only CPR; Chest compression CPR
MeSH Terms: conditions — Heart Arrest; Out-of-Hospital Cardiac Arrest

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CO-CPR Bystander (Experimental): Instructions by dispatcher to trained bystander to provide CPR with chest-compressions only
  Interventions: Procedure: CO-CPR
- S-CPR Bystander (Active Comparator): Instructions by dispatcher to trained bystander to provide CPR with chest-compressions and rescue breaths in a 30:2 ratio
  Interventions: Procedure: S-CPR

INTERVENTIONS:
Procedure: CO-CPR — CPR provided by bystander with chest-compressions only
  Other Names: Compression only CPR; Continous Chest Compressions
  Arms: CO-CPR Bystander
Procedure: S-CPR — CPR with Chest Compressions and Rescue Breaths in a ratio of 30:2
  Other Names: Standard CPR
  Arms: S-CPR Bystander

SUMMARY:
Out-of-hospital cardiac arrest (OHCA) is one of the leading causes of mortality in the industrialized world. Bystander CPR before arrival of the Emergency Medical Service (EMS) is a positive predictor of survival. During the last decade, the best form of bystander CPR has been debated. Chest Compression Only CPR (CO-CPR) has been advocated as a preferable method in situations where the bystander has no previous knowledge in CPR, both because its believed to be equally efficient but also a simplified form of CPR that could lead to a higher incidence of bystander-CPR.

The purpose of this study is to perform av run-in period with focus on safety and feasibility prior to the launch of a larger randomized trial which has a primary end-point of survival. This study will compare OHCA with standard CPR (S-CPR; chest compressions and rescue breaths in a 30:2 fashion) compared to CO-CPR.

DETAILED DESCRIPTION:
Witnessed cases of OHCA with a non-asphyctic aetiology will be the principal study population. According to current guidelines an unresponsive patient with no or agonal breathing is treated as a suspected case of OHCA at the dispatch centre. These cases are eligible for screening for inclusion. If the case is witnessed, the bystander has previous knowledge in CPR and no exclusion criteria are present, the case can be included in the study.

The intervention consists of instructions from a dispatcher at the dispatch centre to bystanders to perform either CO-CPR (intervention) or S-CPR (control).

Instructions to bystanders on how to perform CO-CPR consists of continuous chest compressions without interruptions or rescue breaths. The instructions on how to perform S-CPR in the control group include information on giving chest compressions and rescue breaths in a 30:2 ratio (like current CPR recommendation state).

This is a national study were all dispatch centers in Sweden participate.

The overall study project is conducted in three different phases:

1. Pre study RUN-IN period, for establishing logistical and technical study procedures (completed)
2. PILOT STUDY, with focus feasibility, logistics and safety (Active, not recruting)
3. MAIN STUDY will focus on 30 days survival (primary end point) and other important clinical outcomes (secondary outcomes)

Objective pre study RUN-IN period:

In order to test the technical inclusion procedures, logistics, feasibility and data collection a pre-study RUN-IN period started in Stockholm during 2015.

Objective PILOT study:

The aim of the PILOT study is to assess safety and feasibility of the TANGO2 trial design, as well as intermediate clinical outcomes. The TANGO2 trial started recruitment of patients on January 1st 2017 and last patient was included on December 31st 2018. All patients from the PILOT study will be included in the MAIN STUDY in a seamless design.

Objective MAIN study:

The aim of the MAIN study is to evaluate whether survival to 30 days following instructions to perform CO-CPR is non-inferior compared to instructions to perform S-CPR bystanders in witnessed OHCA where the bystander has previous CPR training. Secondary and exploratory objectives include the evaluation of neurological favorable survival, return of spontaneous circulation, admission to hospital, long-term survival and other clinical outcome variables as well as evaluations of 30-day survival between CO-CPR and S-CPR in pre-specified subgroups. The MAIN study will include patients from the PILOT phase in a seamless design

Experiences from the pre study RUN-IN period and implications for the PILOT and MAIN studies:

The pre-study RUN-IN period started in Stockholm County in 2015 and analysis were performed during 2016. After continuous technological adjustments, the randomization module was integrated within the computer aided dispatch system and was found to functioned well in the end of 2016. However, during pre-study RUN-IN period, one major obstacle was identified. Due to unexpected technological matters and an unanticipated new organization of the dispatch centers in Sweden only about 15% of the cardiac arrest calls for patients suffering cardiac arrest in Stockholm were actually answered by dispatchers in Stockholm; all other calls were transferred to other dispatch centers throughout Sweden. This meant that the dispatchers had to consider the geographical site of the suspected cardiac arrest and remember if that area was part of the study area. This new organization and logistics, were the call could be made in one area and answered and handled at another site and county during the pre-study RUN-IN period, resulted in a far greatly slower inclusion rate than anticipated and made a correct follow-up of patients unmanageable and unreliable. This made it impossible to conduct a PILOT study in Stockholm only.

As a consequence, a decision was made by the steering committee:

A) To move the start of the PILOT study forward, until completion of the national expansion of the study and not to start inclusion of patients into the PILOT study before January 1st 2017. The new length of the PILOT study was set to two years to assure sufficient inclusion of patients to assess safety in terms of survival to hospital admission.

B) That the PILOT study seamlessly will move on into the MAIN study in an inferentially seamless manner after the PILOT phase inclusion ended on Dec 31 2018. This means that patients from the PILOT study will also be included in the MAIN survival study. The outcomes for the PILOT study were changed to not interfere with the primary endpoint of the main survival study (30-day survival).

Inclusion and Exclusion criteria remained unchanged throughout the TANGO2-project.

ELIGIBILITY:
Inclusion Criteria:

* Unconsciousness with no, abnormal or agonal breathing (suspected OHCA)
* The suspected OHCA is witnessed (seen or heard)
* Bystander has previous training in CPR

Exclusion Criteria:

* Age 18 or younger
* Collapse is not witnessed
* Bystander has never been trained in CPR (these bystanders should be instructed to administer CO-CPR in accordance to guidelines).
* Obvious asphyxia, i.e. drowning, strangulation, hanging
* Obvious intoxication or drug overdose
* Pregnancy
* Obvious pregnancy
* Trauma
* Bystander is unwilling to participate or to perform CPR

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1250 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Descriptive measurement of feasibility | 6 months
  * Evaluation of automated inclusion and randomization
  * Evaluation of information of allocation to bystander
  * Adherence to the two protocol, bystanders (S-CPR/CO-CPR)
  * Validation of data collection and sources (please see appendix)
  * Sufficient inclusion of all OHCA during the RUN-IN study period
Descriptive measurement of safety (delay CPR) | 6 months
  * Delay to start of CPR due to screening for inclusion, exclusion, randomization and instructions to the witnesses (S-CPR/CO-CPR)
  * Correct inclusion
  * Correct exclusion
  * Proportion of patients correctly identified as cardiac arrests

SECONDARY OUTCOMES:
Proportions of patients with ventricular fibrillation/ ventricular tachycardia (ITT and PP) | within minutes from arrival of the EMS (day 1)
  Proportions of patients with ventricular fibrillation/ventricular tachycardia at first rhythm analysis
Proportion of patients who achieve return of spontaneous circulation (ROSC) | day 1
  Proportion of patients who achieve return of spontaneous circulation (ROSC)
Survival to hospital admission | day 1
  Survival to hospital admission

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Hollenberg, MD, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Stockholm, Sweden, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No
Data will be published on group level only

REFERENCES:
- [Derived] Riva G, Boberg E, Ringh M, Jonsson M, Claesson A, Nord A, Rubertsson S, Blomberg H, Nordberg P, Forsberg S, Rosenqvist M, Svensson L, Andrell C, Herlitz J, Hollenberg J. Compression-Only or Standard Cardiopulmonary Resuscitation for Trained Laypersons in Out-of-Hospital Cardiac Arrest: A Nationwide Randomized Trial in Sweden. Circ Cardiovasc Qual Outcomes. 2024 Mar;17(3):e010027. doi: 10.1161/CIRCOUTCOMES.122.010027. Epub 2024 Mar 6. PMID 38445487

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-15): https://cdn.clinicaltrials.gov/large-docs/33/NCT02401633/Prot_SAP_001.pdf